CLINICAL TRIAL: NCT06283277
Title: Fetal Clavicular Measurement to Predict Fetal Macrosomia: A Prospective Cohort Study
Brief Title: Fetal Clavicular Measurement to Predict Fetal Macrosomia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mustafa Attyia, principal investigator, Assiut University
Other Study IDs: fetal macrosomia
Record Dates: First submitted 2024-02-04; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Macrosomia, Fetal; Large for Gestational Age; Shoulder Dystocia
Keywords: macrosomia; Hadlock; clavicle; large for gestational age; LGA; clavicle measurement; Youssef's formula; biacromial diameter; estimated fetal weight.; EFW; ultrasound
MeSH Terms: conditions — Fetal Macrosomia; Shoulder Dystocia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Singleton pregnant women at gestational age between 37-42 weeks: estimated fetal weight measured by ultrasound using Hadlock IV formula and Youssef's formula compared with the sensitivity of fetal clavicular measurement.
  Interventions: Device: Obstetric Ultrasound

INTERVENTIONS:
Device: Obstetric Ultrasound — Measuring fetal clavicular length and estimated fetal weight using Hadlock IV formula and Youssef's formula.

SUMMARY:
Macrosomia is associated with increased risks for both the mother and the baby, including complications during delivery, injuries, and even death. The accurate diagnosis of macrosomia is often difficult before birth. There are a number of factors that can increase the risk of macrosomia, such as maternal obesity, diabetes, and excessive weight gain during pregnancy. There are also a number of different techniques that can be used to try to predict macrosomia, but none of them are perfect.

The aim of this study is to evaluate sensitivity of measuring fetal clavicle length in third trimester compared with biacromial diameter and Hadlock formula IV for prediction of fetal macrosomia.

DETAILED DESCRIPTION:
Two terms are applied for fetal overgrowth, Large for gestational age (LGA) meaning fetal birth weight (BW) more than 90th percentile for specific gestational age while macrosomia is an absolute value regardless of gestational age which historically defined as 4000-4500 gm. Those two groups have increased risks for neonatal and maternal complications compared to general population and increase sharply when BW >4500gm, the risks of macrosomia are continuum without threshold defining safe and risky outcome, some authors classify macrosomia into 3 grades, grade 1 (4000gm-4499gm), grade 2(4500-4999), grade 3 (≥5000gm).

Despite its implications, the accurate diagnosis is after birth and its prenatal prediction is poor although published formulas for estimating fetal weight shows correlation with BW, however the variability of the estimate is up to 20% with most of formulas, meta-analysis of 29 studies showed sensitivity of 56% and specificity of 92% in predicting BW ≥ 4000gm accuracy of ultrasound decreases with increasing BW, BW>4500 accurate prediction is only 33-44 % of cases. Given the poor predictability of macrosomia, variety of other techniques and formulas are investigated, neither repeated US examination nor growth curves improves predictability, Youssef's formula measuring biacromial diameter (distance by between both acromial processes which joins clavicles at acromioclavicular joints) and macrosomic specific formula seems to be predictive. In study evaluating clavicle length for shoulder dystocia, it found that measuring clavicle was significant for macrosomia however the limitation is small sample size and its comparison with other fetal biometrics may be needed.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Gestational age between 37-42 weeks.
* Accepting to be included in the study.

Exclusion Criteria:

* Congenital fetal malformation affecting birth weight or affecting clavicle.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women with gestational age between 37 weeks and 42 weeks
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Third trimester clavicle length measurement | 37-42 weeks of gestation
  Sensitivity of third trimester clavicle length measurement in comparison with biacromial diameter and Hadlock IV formula in predicting fetal macrosomia

SECONDARY OUTCOMES:
Establish the relationship between third-trimester clavicle length and shoulder dystocia | Immediately after delivery - postprocedure
  establishing if clavicle length is predictive of shoulder dystocia or not.
Mode of delivery | At the day of delivery
  either vaginal delivery or Cesarean section
Gestational age at the time of delivery. | At the day of delivery
  gestational age and its relation to birth weight
Neonatal Apgar score. | postpartum with 1 and 5 minutes
  neonatal health evaluation
Neonatal bi-acromial diameter | postpartum within 1 to 5 minutes
  measuring actual neonatal biacromial diameter after delivery and its comparision with ultrasound measured biacromial diameter.
Neonatal birth weight | postpartum within 1 to 5 minutes
  neonatal nurse measuring actual neonatal birth weght in grams using digital scale.
Neonatal need for NICU | postpartum within 1 minutes to 5 minutes
  need for neonatal ICU
Neonatal actual clavicle length | postpartum within 1 minutes to 5 minutes
  measuring actual neonatal clavicle length and its comparison with third trimester ultrasound clavicular measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa ElDin Abdelhamid Yusef Hasan, Study Director — Emeritus Professor of obstetrics and gynecology; Ahmed Mohamed Abbas Sobh, Study Director — Assistant Professor of obstetrics and gynecology; Mohamed Mahmoud Abdallah Mahmoud, Study Director — Lecturer of obstetrics and gynecology

REFERENCES:
- [Background] Barth WH, Jackson R. ACOG PRACTICE BULLETIN Clinical Management Guidelines for Obstetrician-Gynecologists. American collage of obstetricians and gynocologists [Internet]. 2020 Jan;135:18-35. Available from: http://journals.lww.com/greenjournal
- [Background] Nesbitt TS, Gilbert WM, Herrchen B. Shoulder dystocia and associated risk factors with macrosomic infants born in California. Am J Obstet Gynecol. 1998 Aug;179(2):476-80. doi: 10.1016/s0002-9378(98)70382-5. PMID 9731856
- [Background] Boulet SL, Alexander GR, Salihu HM, Pass M. Macrosomic births in the united states: determinants, outcomes, and proposed grades of risk. Am J Obstet Gynecol. 2003 May;188(5):1372-8. doi: 10.1067/mob.2003.302. PMID 12748514
- [Background] Zhang X, Decker A, Platt RW, Kramer MS. How big is too big? The perinatal consequences of fetal macrosomia. Am J Obstet Gynecol. 2008 May;198(5):517.e1-6. doi: 10.1016/j.ajog.2007.12.005. PMID 18455528
- [Background] Doty MS, Chen HY, Sibai BM, Chauhan SP. Maternal and Neonatal Morbidity Associated With Early Term Delivery of Large-for-Gestational-Age But Nonmacrosomic Neonates. Obstet Gynecol. 2019 Jun;133(6):1160-1166. doi: 10.1097/AOG.0000000000003285. PMID 31135729
- [Background] Hadlock FP, Deter RL, Harrist RB, Park SK. Estimating fetal age: computer-assisted analysis of multiple fetal growth parameters. Radiology. 1984 Aug;152(2):497-501. doi: 10.1148/radiology.152.2.6739822.
- [Background] Malin GL, Bugg GJ, Takwoingi Y, Thornton JG, Jones NW. Antenatal magnetic resonance imaging versus ultrasound for predicting neonatal macrosomia: a systematic review and meta-analysis. BJOG. 2016 Jan;123(1):77-88. doi: 10.1111/1471-0528.13517. Epub 2015 Jul 29. PMID 26224221
- [Background] Scioscia M, Vimercati A, Ceci O, Vicino M, Selvaggi LE. Estimation of birth weight by two-dimensional ultrasonography: a critical appraisal of its accuracy. Obstet Gynecol. 2008 Jan;111(1):57-65. doi: 10.1097/01.AOG.0000296656.81143.e6. PMID 18165393
- [Background] Zafman KB, Bergh E, Fox NS. Accuracy of sonographic estimated fetal weight in suspected macrosomia: the likelihood of overestimating and underestimating the true birthweight. J Matern Fetal Neonatal Med. 2020 Mar;33(6):967-972. doi: 10.1080/14767058.2018.1511697. Epub 2018 Sep 3. PMID 30099910
- [Background] Sandmire HF. Whither ultrasonic prediction of fetal macrosomia? Obstet Gynecol. 1993 Nov;82(5):860-2. PMID 8414339
- [Background] Aviram A, Yogev Y, Ashwal E, Hiersch L, Danon D, Hadar E, Gabbay-Benziv R. Different formulas, different thresholds and different performance-the prediction of macrosomia by ultrasound. J Perinatol. 2017 Dec;37(12):1285-1291. doi: 10.1038/jp.2017.134. Epub 2017 Sep 14. PMID 28906497
- [Background] Zhang J, Kim S, Grewal J, Albert PS. Predicting large fetuses at birth: do multiple ultrasound examinations and longitudinal statistical modelling improve prediction? Paediatr Perinat Epidemiol. 2012 May;26(3):199-207. doi: 10.1111/j.1365-3016.2012.01261.x. Epub 2012 Feb 10. PMID 22471679
- [Background] Costantine MM, Mele L, Landon MB, Spong CY, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Caritis SN, Sorokin Y, Peaceman AM, Tolosa JE, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network, Bethesda, Maryland. Customized versus population approach for evaluation of fetal overgrowth. Am J Perinatol. 2013 Aug;30(7):565-72. doi: 10.1055/s-0032-1329188. Epub 2012 Nov 12. PMID 23147078
- [Background] Youssef AEA, Amin AF, Khalaf M, Khalaf MS, Ali MK, Abbas AM. Fetal biacromial diameter as a new ultrasound measure for prediction of macrosomia in term pregnancy: a prospective observational study. J Matern Fetal Neonatal Med. 2019 Aug;32(16):2674-2679. doi: 10.1080/14767058.2018.1445714. Epub 2018 Mar 7. PMID 29478363
- [Background] Porter B, Neely C, Szychowski J, Owen J. Ultrasonographic Fetal Weight Estimation: Should Macrosomia-Specific Formulas Be Utilized? Am J Perinatol. 2015 Aug;32(10):968-72. doi: 10.1055/s-0035-1545664. Epub 2015 Mar 2. PMID 25730134
- [Background] Terzi E. A new approach to predicting shoulder dystocia: fetal clavicle measurement. Turk J Med Sci. 2021 Aug 30;51(4):1932-1939. doi: 10.3906/sag-2011-145. PMID 33843172
- [Background] Yarkoni S, Schmidt W, Jeanty P, Reece EA, Hobbins JC. Clavicular measurement: a new biometric parameter for fetal evaluation. J Ultrasound Med. 1985 Sep;4(9):467-70. doi: 10.7863/jum.1985.4.9.467. PMID 3903198
- [Background] Sherer DM, Sokolovski M, Dalloul M, Khoury-Collado F, Osho JA, Lamarque MD, Abulafia O. Fetal clavicle length throughout gestation: a nomogram. Ultrasound Obstet Gynecol. 2006 Mar;27(3):306-10. doi: 10.1002/uog.2706. PMID 16450360
- [Background] Shmueli A, Salman L, Hadar E, Aviram A, Bardin R, Ashwal E, Gabbay-Benziv R. Sonographic prediction of macrosomia in pregnancies complicated by maternal diabetes: finding the best formula. Arch Gynecol Obstet. 2019 Jan;299(1):97-103. doi: 10.1007/s00404-018-4934-y. Epub 2018 Oct 16. PMID 30327863